CLINICAL TRIAL: NCT03121131
Title: How Important is a Clinical Data for a Radiologist? A Double-Blinded Randomized Controlled Trial of Radiologic Interpretation of Ventral Hernias Following Selectively-Provided Clinical Information
Brief Title: CT and Radiologist RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mike K Liang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSC-MS-17-0277
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Accurate Clinical Exam Findings (Other): Radiologists will be provided with accurate clinical exam data.
  Interventions: Other: Clinical Exam Findings
- Inaccurate Clinical Exam Findings (Other): Radiologists will be provided with purposefully incorrect clinical exam data
  Interventions: Other: Inaccurate Clinical Exam Findings
- No Clinical Exam Findings (Other): Radiologists will be not be provided with any clinical exam data
  Interventions: Other: No clinical exam findings

INTERVENTIONS:
Other: Clinical Exam Findings — Findings found on clinical exam of a patient the radiologist will be reading CT scans of.
  Arms: Accurate Clinical Exam Findings
Other: Inaccurate Clinical Exam Findings — Inaccurate findings are given to the radiologists
  Arms: Inaccurate Clinical Exam Findings
Other: No clinical exam findings — No clinical exam findings are given to the radiologists
  Arms: No Clinical Exam Findings

SUMMARY:
The use of computed tomography (CT) imaging is rapidly increasing in healthcare. Despite physicians' growing reliance on radiological assessments, however, the reliability and accuracy of reads are highly variable. Inconsistencies may result from multiple factors.

The researchers hypothesize that the presence and quality of clinical information will affect radiologist's assessment of CT scans for the presence/absence of a ventral hernia.

ELIGIBILITY:
Participants are radiologists at LBJ Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Hernia detected on CT | CT taken within 1 year
  proportion of hernias detected on CT

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health at Lyndon B. Johnson General Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Cherla DV, Bernardi K, Blair KJ, Chua SS, Hasapes JP, Kao LS, Ko TC, Matta EJ, Moses ML, Shiralkar KG, Surabhi VR, Tammisetti VS, Viso CP, Liang MK. Importance of the physical exam: double-blind randomized controlled trial of radiologic interpretation of ventral hernias after selective clinical information. Hernia. 2019 Oct;23(5):987-994. doi: 10.1007/s10029-018-1856-3. Epub 2018 Nov 14. PMID 30430273